CLINICAL TRIAL: NCT06477081
Title: Keratorefractive Lenticule Extraction (KLEx) Versus Femtosecond Laser-assisted in Situ Keratomileusis (FS-LASIK) for the Treatment of Myopia and Compound Myopic Astigmatism
Brief Title: KLEx Versus FS-LASIK for the Treatment of Myopia and Compound Myopic Astigmatism
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Oftalmología Fundación Conde de Valenciana (Other)
Responsible Party: Principal Investigator, Nicolas Kahuam Lopez, Consultant, Instituto de Oftalmología Fundación Conde de Valenciana
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CI-017-2024
Record Dates: First submitted 2024-06-17; First posted 2024-06-27 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Myopia; Astigmatism; Myopic Astigmatism
Keywords: KLEx; LASIK; FS-LASIK; Refractive Surgery; Astigmatism; Myopia
MeSH Terms: conditions — Myopia; Astigmatism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Allocation sequence concealment will be done with sealed opaque envelopes. The envelope will be open prior to the intervention only to surgical team. The technique will not be known by the patient or the staff responsible of the follow-up.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FemtoLASIK (Active Comparator): For the FS-LASIK technique, the following steps will be followed: application of topical anesthesia to mitigate discomfort and pain throughout the procedure, and the patient will be covered with a sterile drape. Subsequently, the patient will be aligned to artificially flatten the entire corneal surface, ensuring head stability with a slight tilt to optimize surgical access and avoid nasal interference. The femtosecond laser system use will be the ATOS operating system (Schwind eye-tech-solutions, Mainparkstraße 6-10, 63801 Kleinostheim, Germany), which is responsible for creating a corneal incision to create the flap, with controlled precision to ensure proper separation of corneal layers. The excimer laser will be the Amaris (Schwind eye-tech-solutions, Mainparkstraße 6-10, 63801 Kleinostheim, Germany), responsible for performing refractive correction on the cornea through selective photoablation. Following photoablation, the flap will be carefully repositioned, and upon completion
  Interventions: Procedure: FS-LASIK procedure
- Keratorefractive lenticule extraction (Active Comparator): For the KLEx technique, the following steps will be followed: after topical anesthesia, a sterile drape is placed over the patient, and a speculum is inserted into the eye, centered, and aligned with a curved interface cone before applying suction. The laser used will be the ATOS operating system (Schwind eye-tech-solutions, Mainparkstraße 6-10, 63801 Kleinostheim, Germany), which performs photo-dissection starting from the posterior surface of the refractive lenticule, followed by the creation of the lenticule edge. The anterior surface of the refractive lenticule is formed by extending beyond the posterior diameter of the lenticule by 0.5 mm to form the anterior flap, followed by a peripheral cut. Specific FS laser parameters are employed for each patient. Subsequently, the suction is released, and a Siebel spatula is used to separate and reflect the flap. Finally, the refractive lenticule is extracted using toothless forceps through the small incision. Once the procedure is complet
  Interventions: Procedure: KLEx

INTERVENTIONS:
Procedure: FS-LASIK procedure — For the FS-LASIK technique, the following steps will be followed: application of topical anesthesia to mitigate discomfort and pain throughout the procedure, and the patient will be covered with a sterile drape. Subsequently, the patient will be aligned to artificially flatten the entire corneal surface, ensuring head stability with a slight tilt to optimize surgical access and avoid nasal interference. The femtosecond laser system use will be the ATOS operating system (Schwind eye-tech-solutions, Mainparkstraße 6-10, 63801 Kleinostheim, Germany), which is responsible for creating a corneal incision to create the flap, with controlled precision to ensure proper separation of corneal layers. The excimer laser will be the Amaris (Schwind eye-tech-solutions, Mainparkstraße 6-10, 63801 Kleinostheim, Germany), responsible for performing refractive correction on the cornea through selective photoablation. Following photoablation, the flap will be carefully repositioned, and upon completion o
  Arms: FemtoLASIK
Procedure: KLEx — For the KLEx technique, the following steps will be followed: after topical anesthesia, a sterile drape is placed over the patient, and a speculum is inserted into the eye, centered, and aligned with a curved interface cone before applying suction. The laser used will be the ATOS operating system (Schwind eye-tech-solutions, Mainparkstraße 6-10, 63801 Kleinostheim, Germany), which performs photo-dissection starting from the posterior surface of the refractive lenticule, followed by the creation of the lenticule edge. The anterior surface of the refractive lenticule is formed by extending beyond the posterior diameter of the lenticule by 0.5 mm to form the anterior flap, followed by a peripheral cut. Specific FS laser parameters are employed for each patient. Subsequently, the suction is released, and a Siebel spatula is used to separate and reflect the flap. Finally, the refractive lenticule is extracted using toothless forceps through the small incision. Once the procedure is complete
  Arms: Keratorefractive lenticule extraction

SUMMARY:
FemtoLASIK is a type of laser eye surgery used to correct vision problems such as nearsightedness, farsightedness, and astigmatism. It involves two main steps: creating a flap and reshaping the cornea. Refractive lenticule extraction, (KLEx) is another laser eye surgery method to correct vision issues, which involves creating and extracting a lenticule without the need of a flap. The investigators will evaluate and compare the efficacy and safety of these two procedures.

DETAILED DESCRIPTION:
Keratorefractive lenticule extraction (KLEx) is a refractive surgery technique that does not require the creation of a flap to correct the defects. The potential advantages of this technique are related to the absence of a flap, which could make it the gold standard of refractive surgery. On the other hand, femtosecond-assisted laser in-situ keratomileusis (FS-LASIK) is the most widely practiced refractive surgery worldwide, as it offers excellent visual outcomes but does require the creation of a flap to correct the defects. The objective of this study is to evaluate the effectiveness and safety of KLEx versus FS-LASIK as a treatment option in patients with myopia or compound myopic astigmatism. This is a prospective randomized study. A total of 80 participants will be randomized into two groups, the KLEx group and FS-LASIK group. Following randomization, participants will be followed on the first day after the surgery, 1 week, 1, 3, 6, and 12 months. The primary outcome is the refractive predictability at every postoperative point after surgery, which is the proportion of the number of eyes achieving a postoperative spherical equivalent within ± 0.5 diopters of the intended target. Secondary outcome parameters include quality vision measurements, refraction, visual acuity, and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 years or older
* Corneal tomography without alterations
* Myopia between -0.50 and -12.00 D
* Astigmatism between -0.50 and -6.00 D

Exclusion Criteria:

* Previous eye surgeries
* Pregnancy
* Progressive or unstable myopia and/or compound myopic astigmatism
* Ocular surface disease

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Uncorrected Visual Acuity | Day 1, week 1, months 1, 3, 6 & 12th after surgery.
  Visual acuity without correction after surgery.

SECONDARY OUTCOMES:
Postoperative spherical equivalent | Day 1, week 1, months 1, 3, 6 & 12th after surgery.
  Overall refractive power that has both spherical and cylindrical components.
Corrected Distance Visual Acuity | Day 1, week 1, months 1, 3, 6 & 12th after surgery.
  Visual acuity after surgery with refractive correction
Loss of 2 or more lines of BCVA | Day 1, week 1, months 1, 3, 6 & 12th after surgery.
  Loss of 2 or more lines of best corrected visual acuity
Eyes with 0.5 Diopters within refractive target. | Day 1, week 1, months 1, 3, 6 & 12th after surgery.
  Proportion of eye within 0.5 Diopters of refactive target.

OTHER OUTCOMES:
Adverse events. | Through study completion, an average of 1 year
  Dry eye, haze, flap complications, diffuse lamellar keratitis, corneal ectasia, epithelial ingrowth, or any other adverse event.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto de Oftalmología Conde de Valenciana, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pradhan KR, Arba Mosquera S. SmartSight Correction of Compound Myopic Astigmatism Treatments With Preoperative Astigmatism > 1.00 Diopter Using the SCHWIND ATOS: A Retrospective Case Series. J Refract Surg. 2024 May;40(5):e328-e335. doi: 10.3928/1081597X-20240415-02. Epub 2024 May 1. PMID 38717080
- [Background] Igras E, Czarnota-Nowakowska B, O'Caoimh R. Comparison of the Clinical Effectiveness of Correcting Different Types of Astigmatism with Small Incision Lenticule Extraction. J Clin Med. 2023 Nov 6;12(21):6941. doi: 10.3390/jcm12216941. PMID 37959406
- [Background] Foo VHX, Liu YC, Ang M, Htoon HM, Ting DSJ, Mehta JS. Comparative Study of Primary SMILE, SMILE Enhancement, and Femtosecond Laser-Assisted LASIK on Higher Order Aberrations and Corneal Densitometry. J Refract Surg. 2024 May;40(5):e291-e303. doi: 10.3928/1081597X-20240314-01. Epub 2024 May 1. PMID 38717083
- [Derived] Muleiro-Alvarez M, Vera-Duarte GR, Medina-Estrada EA, Ortiz-Morales G, Ramirez-Miranda A, Navas A, Graue-Wiechers EL, Graue-Hernandez EO, Kahuam-Lopez N. Keratorefractive lenticule extraction (KLEx) versus femtosecond laser-assisted in situ keratomileusis (FS-LASIK) for the treatment of myopia and compound myopic astigmatism: study protocol of a randomised clinical trial in Mexico. BMJ Open. 2025 Dec 23;15(12):e097192. doi: 10.1136/bmjopen-2024-097192. PMID 41436254